CLINICAL TRIAL: NCT00274339
Title: A Comparison of Prevacid 30mg BID Plus Lifestyle Modifications Versus Lifestyle Modifications Alone for the Treatment of Laryngopharyngeal Reflux (LPR) in Adults
Brief Title: Prevacid vs Lifestyle Modifications for the Treatment of LPR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hodge, Kenneth M., M.D. (Individual)
Collaborators: TAP Pharmaceutical Products Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LPR-04-01
Record Dates: First submitted 2006-01-06; First posted 2006-01-10 (Estimated); Last update posted 2007-06-25 (Estimated); Status verified 2007-06

CONDITIONS: Laryngopharyngeal Reflux
Keywords: Laryngopharyngeal Reflux; Prevacid; Lifestyle changes; Reflux Finding Score; Reflux Symptom Index; Laryngoscopy
MeSH Terms: conditions — Laryngopharyngeal Reflux | interventions — Lansoprazole; BID protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Prevacid 30mg BID
Behavioral: Lifestyle changes of exercise and diet changes for weight loss and avoidance of reflux inducing foods.

SUMMARY:
The purpose of this study is to evaluate changes in scores on the Reflux Finding Score and Reflux Symptom Index over a 24 week period. To enroll subjects must score at least a 13 on the Reflux Symptom Index and at least a 5 on the Reflux Finding Score. All subjects will receive education on lifestyle modifications with a nutritionist and exercise trainer. All subjects will be expected to comply with lifestyle modifications for the entire study period of 24 weeks. Half of all subjects will receive Prevacid 30mg BID and half will receive placebo BID for 24 weeks. Subjects will have 4 office visits over 24 weeks and weekly contacts with the study staff to assess Reflux Symptom Index and any health or medication changes.

DETAILED DESCRIPTION:
The results of studies evaluating PPI therapy versus lifestyle modifications for the treatment of LPR have not been conclusive. However, many of these studies were conducted at tertiary care centers. We will look at patients presenting with LPR symptoms in a community setting. All subjects will have an exam of their larynx via laryngoscopy at each of the 4 study visits (screening, week 6, week 12, and week 24). Based on exam findings, the physician will complete the Reflux Finding Score. The subjects will also complete the Reflux Symptom Index weekly to assess for changes in their symptoms. The statistical analysis of this study will include evaluating changes in the Reflux Finding Scores and Reflux Symptom Index scores over the 24 weeks of study participation.

ELIGIBILITY:
Inclusion Criteria:

Symptoms of LPR for at least one month, Score of 5 or greater on Reflux Finding Score, Score of 13 or greater on Reflux Symptom Index, and Willing to follow lifestyle modifications.

Exclusion Criteria:

Currently taking PPI twice daily for the treatment of LPR, Women who are pregnant or lactating, History of duodenal or gastric ulcer in the past 5 years, erosive esophagitis, or esophageal obstruction, History of any hypersecretory condition, History of Barrett's esophagus, History of hematemesis in the past 6 months, Currently taking ketoconazole, digoxin, Iron, ampicillin, theophylline, warfarin, or sucralfate, or Suspected disease of the larynx not related to LPR.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Estimated)
Dates: Start 2005-12; Study Completion 2008-06 (Estimated)

PRIMARY OUTCOMES:
To compare the numbers of subjects with a Reflux Symptom Index score of less than 13 at visit 3 | 6 months

SECONDARY OUTCOMES:
To evaluate the changes in Reflux Finding Score and Reflux Symptom Index from initial scores at screening to final assessment at visit 3. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth M Hodge, MD, Principal Investigator — Commonwealth Ear, Nose & Throat
Locations (1):
- Commonwealth Ear, Nose & Throat, Louisville, Kentucky, United States

REFERENCES:
- [Background] Belafsky PC, Postma GN, Koufman JA. Validity and reliability of the reflux symptom index (RSI). J Voice. 2002 Jun;16(2):274-7. doi: 10.1016/s0892-1997(02)00097-8. PMID 12150380
- [Background] Belafsky PC, Postma GN, Koufman JA. The validity and reliability of the reflux finding score (RFS). Laryngoscope. 2001 Aug;111(8):1313-7. doi: 10.1097/00005537-200108000-00001. PMID 11568561
- [Background] Belafsky PC, Postma GN, Amin MR, Koufman JA. Symptoms and findings of laryngopharyngeal reflux. Ear Nose Throat J. 2002 Sep;81(9 Suppl 2):10-3. PMID 12353425
- [Background] Cohen JT, Bach KK, Postma GN, Koufman JA. Clinical manifestations of laryngopharyngeal reflux. Ear Nose Throat J. 2002 Sep;81(9 Suppl 2):19-23. PMID 12353427
- [Background] Koufman JA. Laryngopharyngeal reflux 2002: a new paradigm of airway disease. Ear Nose Throat J. 2002 Sep;81(9 Suppl 2):2-6. PMID 12353428
- [Background] Koufman JA. Laryngopharyngeal reflux is different from classic gastroesophageal reflux disease. Ear Nose Throat J. 2002 Sep;81(9 Suppl 2):7-9. PMID 12353431
- [Background] Postma GN, Belafsky PC, Aviv JE, Koufman JA. Laryngopharyngeal reflux testing. Ear Nose Throat J. 2002 Sep;81(9 Suppl 2):14-8. PMID 12353426
- [Background] Postma GN, Johnson LF, Koufman JA. Treatment of laryngopharyngeal reflux. Ear Nose Throat J. 2002 Sep;81(9 Suppl 2):24-6. PMID 12353429
- [Background] Vaezy, M & Postma, GN. Laryngopharyngeal Reflux from an ENT and GI Perspective Course. October 21, 2004. Louisville, KY.